CLINICAL TRIAL: NCT06798584
Title: Rough Journey to Menopause: How Does Perimenopausal Menorrhagia Affect Women's Quality of Life and Cognitive Function?
Brief Title: How Does Perimenopausal Menorrhagia Affect Women's Quality of Life and Cognitive Function?
Acronym: MENO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Laura Murray Kolb, Professor & Department Head, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2024-506
Record Dates: First submitted 2024-11-15; First posted 2025-01-29 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Iron Deficiency Anemia Treatment; Iron Deficiency; Iron Deficiency (Without Anemia)
Keywords: Iron; Perimenopause; Iron Deficiency Anemia; Iron Deficiency; Cognitive Function; Quality of Life; Mood; Quality of Family Relationships; Menopause; Perimenopausal Menorrhagia; Abnormal Uterine Bleeding; Menopause Transition; Women's Health
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency; Metrorrhagia

STUDY DESIGN:
Intervention Model Description: Participants will be classified as iron sufficient, iron deficient, or iron deficient anemic according to the following parameters. To be classified as iron deficient anemic (IDA): Hb between 100 and 119 g/L, and at least 2 of the following iron deficiency parameters: mean corpuscular volume (MCV) < 80 fL, transferrin saturation (TSAT) <15%, serum ferritin (Ft) <15 ug/L, serum transferrin receptor >8.3 mg/L, serum hepcidin <8 ng/mL; to be classified as iron deficient without anemia (ID): at least 2 of the abnormal values listed above with a Hb>=120 g/L; to be classified as iron sufficient (IS): Hb >=120 g/L, MCV >80 fL, TSAT >15%, Ft >20 ug/L, TfR < 6 mg/L, and hepcidin >8 ng/mL. Any participant with a Hb <100 g/L will be excluded from the study as being too anemic and be referred to a physician for immediate treatment of the anemia. Any participant with a Ft>200 ug/L will be excluded from the study and advised to follow up with a physician.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Iron Sufficient - Placebo (Placebo Comparator): Women classified as iron sufficient given a 4-month supply of gelatin capsules
  Interventions: Dietary Supplement: 21st Century Gelatin Capsules
- Iron Sufficient - Iron Supplements (Experimental): Women classified as iron sufficient given a 4-month supply of iron supplements
  Interventions: Dietary Supplement: FeoSol Original Iron Supplement Tablets
- Iron Deficient - Placebo (Placebo Comparator): Women classified as iron deficient given a 4-month supply of gelatin capsules
  Interventions: Dietary Supplement: 21st Century Gelatin Capsules
- Iron Deficient - Iron Supplements (Experimental): Women classified as iron deficient given a 4-month supply of iron supplements
  Interventions: Dietary Supplement: FeoSol Original Iron Supplement Tablets
- Iron Deficient (Anemic) - Placebo (Placebo Comparator): Women classified as anemic given a 4-month supply of gelatin capsules
  Interventions: Dietary Supplement: 21st Century Gelatin Capsules
- Iron Deficient (Anemic) - Iron Supplements (Experimental): Women classified as anemic given a 4-month supply of iron supplements
  Interventions: Dietary Supplement: FeoSol Original Iron Supplement Tablets

INTERVENTIONS:
Dietary Supplement: FeoSol Original Iron Supplement Tablets — 325 mg of ferrous sulfate containing 65 mg of elemental iron
  Arms: Iron Deficient (Anemic) - Iron Supplements; Iron Deficient - Iron Supplements; Iron Sufficient - Iron Supplements
Dietary Supplement: 21st Century Gelatin Capsules — 600 mg
  Arms: Iron Deficient (Anemic) - Placebo; Iron Deficient - Placebo; Iron Sufficient - Placebo

SUMMARY:
The goal of this clinical trial is to investigate how iron status and heavy bleeding during the menopausal transition affect women's cognitive function and quality of life. The main questions it aims to answer are:

* What is the association between iron status, cognitive function, mood, quality of family relationships, and quality of life in perimenopausal women?
* How does iron repletion, via supplementation, affect cognitive function, mood, quality of family relationships, and quality of life in perimenopausal women?

The investigators will compare the effect of iron supplements to a placebo (gelatin capsule) to see if iron supplements could improve iron status, cognitive function, mood, quality of family relationships, and quality of life of iron-deficient and/or anemic women undergoing the menopausal transition.

Each participant will:

* Make 2 visits (about 2 hours each - baseline and endline) to the Clinical Research Center at Purdue
* Make a very brief visit at midpoint (about 10 minutes) for a checkup
* Take a daily study supplement or placebo for 4 months

DETAILED DESCRIPTION:
(i) Recruitment: The investigators will recruit participants through advertisements and referrals. The investigators will utilize advertisements in Purdue Today, women's health clinics located in West Lafayette, Lafayette, and Indianapolis, and other social media platforms. Inclusion criteria are: all participants are undergoing natural perimenopause, English-speaking, and in general good health as documented by each woman's personal report that the participant is without any past history of a chronic health condition. The participants who have been using iron supplementation prior to the study may participate if the participants agree to discontinue the use of iron supplementation for the duration of the study. Lastly, individuals taking psychoactive drugs or with a history of hematological disorders will be excluded from the study.

(ii) Screening: Interested participants may either call or email the investigators using contact information found on the flyer or complete a short survey, which can be accessed via QR code on the flyer.

(iii) Randomization to treatment: Once the participants are classified as belonging to the IDA, ID, or IS groups, the participants will then be randomly assigned (within group) to receive either an iron supplement or a placebo for 4 months (previous studies have indicated a significant improvement in iron status and functional outcomes with a 4-month intervention period). FeoSol Original Iron Supplement Tablets (325 mg of ferrous sulfate containing 65 mg of elemental iron) will be used for the treatment (this have used this successfully in past studies) and 21st Century Gelatin Capsules (600 mg) will be used for the placebo (gelatin capsules have been used successfully for the placebo group, in past studies). Participants will be advised to take one capsule/tablet each day with food and store the given treatment out of the reach of children. Weekly phone calls or texts will be placed to each of the participants as a reminder to take supplements and to check tolerance to iron supplements. If intolerance to iron supplements are reported, participants may have an option to stop taking iron supplements. During weekly phone calls or texts, participants will also be asked if participants have started any new medications or become pregnant. If a participant becomes pregnant, participant's participation in the study will be terminated at that time. If a participant's physician is concerned about what the participants may be taking for this study, a participant's physician may contact either Mun Choi or Laura Murray-Kolb, whose contact information will be provided to all participants to share with physicians. Compliance will be measured through pill counts half-way through and at the end of the study. Group and treatment assignment will be blinded to the participants as well as the investigators.

(iv) Assessment of quality of life, mood, and family relationships: Assessment of these variables will take place before the blood draw at the Purdue Clinical Research Center at both baseline and endline of the study. Quality of life will be assessed using the self-administered MOS 36-Item Short Form Health Survey (SF-36) and the Menopause-Specific Quality of Life Questionnaire (MENQOL). These scales have been used extensively and shown to have good reliability with coefficients equal to or greater than 0.80 in most studies. For the assessment of mood, participants will be asked to complete the Beck Depression Inventory-II (BDI-II). The BDI-II is a 21-item self-reporting questionnaire and items will be summed to create a total score with higher scores indicating higher levels of depression. It has been widely used in research and clinical settings to measure depressive symptoms according to the diagnostic criteria listed in the Diagnostic and Statistical Manual for Mental Disorders. The BDI-II has been tested for validity and reliability in different populations and has good internal consistency and reliability. Family relationships will be assessed using the Family Adaptability and Cohesion Evaluation Scale IV Short Form (FACES-IV-SF). Ratio scores that are less than 1 indicate unbalanced families, or lower quality of interactions among family members. A recent validation study showed that the FACES-IV-SF demonstrated adequate reliability and good fit to the data as evidenced by the Cronbach's alphas for the subscales ranging from 0.63 (Enmeshment) to 0.93 (Satisfaction). All family members over the age of 12 (age of 13-17) that live with participants will be asked to complete this questionnaire. For family members who are under the age of 18, parental consent will be obtained when obtaining participant's written consent and youth assent will be obtained before the administration of the FACES-IV questionnaire via Qualtrics. For family members who are at or over the age of 18, individual consent will be obtained before the administration of the FACES-IV questionnaire via Qualtrics.

(v) Computerized measures of cognitive function: Executive function is an umbrella term that is used to describe complex mental operations such as planning, time perception, working memory, inhibition, self-monitoring and regulation, motor control, regulation of emotion, and motivation. To assess multiple domains of executive function in women with perimenopausal menorrhagia, the Psychology Experiment Building Language (PEBL) platform will be utilized to evaluate cognitive domains that were shown to be affected by iron status in previous studies. The PEBL is a software package allowing the creation of computerized tests for experimental use and neuropsychological testing, and has been widely used in different populations to assess cognitive performance. Thus, the following tests will be performed through the PEBL to assess five domains of cognition in perimenopausal women in a lighting and temperature-controlled testing environment:

Berg Card Sorting Test: The short 64-card version of the Berg Card Sorting Test (BCST) will be used as one measure of executive function in women. The test entails sorting cards based on shape, color, or number. A participant is given feedback (correct or incorrect) after each sorting, and participant may need to adjust sorting strategy based on the feedback received. During the test, the sorting rule changes (unbeknownst to the participant) and when it does, a participant must adjust sorting strategy accordingly. The BCST is used to distinguish diminished mental capacity and the shortened 64-card version of the BCST has been validated for use.

Attention Network Task: The Attention Network Task (ANT) is designed to assess three components of executive attention in a 30-minute testing session. The three components of executive attention that the ANT assesses include alerting (the ability to perceive that there is something to be attentive to), orienting (the ability to direct and shift attention to where it is needed), and conflict (the ability to filter out competing information). This test will present a sequence of visual stimuli where a participant will be shown cues in the form of either one or two asterisks in order to predict an upcoming target presentation and/or to orient the target's location. The cue is then followed by the presentation of target arrows, which may appear individually or in an arrangement of five arrows. A participant will be asked to respond by indicating which way the central arrow is facing, and scores for each network of attention will be calculated by reaction time subtractions of different stimulus combinations. The ANT has been performed by different populations and has been validated for use.

Go/No-Go Task: The Go/No-Go (GNG) Task is designed to assess one's ability to inhibit impulsivity while responding to go cues. During the GNG task, a participant is presented with a 2 x 2 pattern with one star in each square. The participant is instructed to follow a sequential presentation of letters and respond to the target letter (P) by pressing a button on the keyboard as quickly as possible, while suppressing responses to the non-target letter (R). The sequential presentation of letters is randomly generated and presented for 500 milliseconds in one of four squares with a 1500-millisecond interstimulus interval.

Tower of London Task: The Tower of London (TOL) Task is designed to assess one's efficiency in planning. During the TOL task, a participant is provided with colored disks that can be placed in three stacks with a maximum height of 1, 2, or 3 disks. Participants need to match a target configuration by moving one disk at a time and trying to do so in as few moves as possible. Prior to the task, practice trials are provided, and participants will be instructed to plan their entire sequence of moves mentally before initiating. The outcomes of this task include excess moves, planning time, and total time.

Sternberg Memory Search Task: The Sternberg Memory Search (SMS) Task is designed to evaluate one's working memory. During the SMS task, a participant is required to remember a series of letters presented one at a time and is then probed about whether particular letters were part of the presented set. In addition to accuracy, the amount of transmitted information, or throughput, will be calculated to correct for chance level [throughput = {(uncorrected overall accuracy - 0.5) / 0.5} x the number of items included in the memory set].

ELIGIBILITY:
Inclusion Criteria:

* Undergoing natural perimenopause
* English-speaking
* In general good health as documented by each woman's personal report that the participant is without any past history of a chronic health condition

Exclusion Criteria:

* Taking psychoactive drugs
* A history of hematological disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Iron Status Assessment | From enrollment to the end of treatment at 4 months
  The investigators will measure plasma iron (mcg/dL).
Iron Status Assessment | From enrollment to the end of treatment at 4 months
  The investigators will measure total iron binding capacity (TIBC) (mcg/dL).
Iron Status Assessment | From enrollment to the end of treatment at 4 months
  The investigators will measure transferrin saturation (TSAT) (%).
Iron Status Assessment | From enrollment to the end of treatment at 4 months
  The investigators will measure serum ferritin (Ft) (μg/L).
Iron Status Assessment | From enrollment to the end of treatment at 4 months
  The investigators will measure serum transferrin receptor (TfR) (mg/L).
Iron Status Assessment | From enrollment to the end of treatment at 4 months
  The investigators will measure CBC parameters (including hemoglobin (Hb) (g/dL), hematocrit (Hct) (%), mean corpuscular volume (MCV) (fL), and red blood cell distribution width (RDW) (fL)), which are measured in whole blood.
Iron Status Assessment | From enrollment to the end of treatment at 4 months
  The investigators will measure serum hepcidin (ng/mL).
Iron Status Assessment | From enrollment to the end of treatment at 4 months
  The investigators will calculate body Fe (mg/kg) using Cook's formula.
Inflammation Assessment | From enrollment to the end of treatment at 4 months
  The investigators will measure α-1-acid glycoprotein (g/L) as an indicator of inflammation. In cases where inflammation is indicated, ferritin (μg/L) and TfR (mg/L) levels will not be used to assess iron status or concentrations will be adjusted using either the Thurnham or BRINDA methods.
Inflammation Assessment | From enrollment to the end of treatment at 4 months
  The investigators will measure C-reactive protein (mg/L) as an indicator of inflammation. In cases where inflammation is indicated, ferritin (μg/L) and TfR (mg/L) levels will not be used to assess iron status or concentrations will be adjusted using either the Thurnham or BRINDA methods.
Cognitive Function Assessment | From enrollment to the end of treatment at 4 months
  To assess multiple domains of executive function, the Psychology Experiment Building Language (PEBL) platform will be utilized to evaluate cognitive domains that were shown to be affected by iron status in previous studies. Berg Card Sorting Test (# of categories completed and # of perseverative errors) will be performed through the PEBL to assess executive function in participants in a lighting and temperature-controlled testing environment.
Cognitive Function Assessment | From enrollment to the end of treatment at 4 months
  To assess multiple domains of executive function, the Psychology Experiment Building Language (PEBL) platform will be utilized to evaluate cognitive domains that were shown to be affected by iron status in previous studies. Attention Network Task (% correct for accuracy and reaction time, alerting, orienting, and conflict measurements in milliseconds) will be performed through the PEBL to assess alerting, orienting, and conflict in participants in a lighting and temperature-controlled testing environment.
Cognitive Function Assessment | From enrollment to the end of treatment at 4 months
  To assess multiple domains of executive function, the Psychology Experiment Building Language (PEBL) platform will be utilized to evaluate cognitive domains that were shown to be affected by iron status in previous studies. Go Task: The Go/No-Go (% correct for accuracy and reaction time in milliseconds) will be performed through the PEBL to assess the ability to inhibit impulsivity while responding to go cues in participants in a lighting and temperature-controlled testing environment.
Cognitive Function Assessment | From enrollment to the end of treatment at 4 months
  To assess multiple domains of executive function, the Psychology Experiment Building Language (PEBL) platform will be utilized to evaluate cognitive domains that were shown to be affected by iron status in previous studies. Tower of London Task (# of excess moves and planning and solution time in milliseconds) will be performed through the PEBL to assess the efficiency in planning in participants in a lighting and temperature-controlled testing environment.
Cognitive Function Assessment | From enrollment to the end of treatment at 4 months
  To assess multiple domains of executive function, the Psychology Experiment Building Language (PEBL) platform will be utilized to evaluate cognitive domains that were shown to be affected by iron status in previous studies. Sternberg Memory Search Task (% correct for accuracy, reaction time in milliseconds, and # of throughput) will be performed through the PEBL to assess working memory in participants in a lighting and temperature-controlled testing environment.
Quality of Life | From enrollment to the end of treatment at 4 months
  Quality of life will be assessed using the self-administered MOS 36-Item Short Form Health Survey (SF-36), with a score ranging from 0 to 100, where higher scores indicate better health.
Quality of Life | From enrollment to the end of treatment at 4 months
  Quality of life will be assessed using the Menopause-Specific Quality of Life Questionnaire (MENQOL), with a score ranging from 0 to 6, where higher scores indicate worse quality of life.
Assessment of Mood | From enrollment to the end of treatment at 4 months
  Mood will be assessed using the Beck Depression Inventory-II (BDI-II) (with a score ranging from 0 to 63, where higher scores indicate worse depressive symptoms).
Assessment of Family Relationships | From enrollment to the end of treatment at 4 months
  Family relationships will be assessed using the Family Adaptability and Cohesion Evaluation Scale IV Short Form (FACES-IV-SF) (with a score ranging from 0-1, where scores less than one represents families with problematic functioning).

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Murray-Kolb, PhD, Principal Investigator — Purdue University
Locations (1):
- Stone Hall, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Whiteley J, DiBonaventura Md, Wagner JS, Alvir J, Shah S. The impact of menopausal symptoms on quality of life, productivity, and economic outcomes. J Womens Health (Larchmt). 2013 Nov;22(11):983-90. doi: 10.1089/jwh.2012.3719. Epub 2013 Oct 1. PMID 24083674
- [Background] Wenger MJ, Murray-Kolb LE, Nevins JE, Venkatramanan S, Reinhart GA, Wesley A, Haas JD. Consumption of a Double-Fortified Salt Affects Perceptual, Attentional, and Mnemonic Functioning in Women in a Randomized Controlled Trial in India. J Nutr. 2017 Dec;147(12):2297-2308. doi: 10.3945/jn.117.251587. Epub 2017 Oct 11. PMID 29021371
- [Background] Wenger MJ, Murray Kolb LE, Scott SP, Boy E, Haas JD. Modeling relationships between iron status, behavior, and brain electrophysiology: evidence from a randomized study involving a biofortified grain in Indian adolescents. BMC Public Health. 2022 Jul 6;22(1):1299. doi: 10.1186/s12889-022-13612-z. PMID 35794587
- [Background] Wenger MJ, DellaValle DM, Murray-Kolb LE, Haas JD. Effect of iron deficiency on simultaneous measures of behavior, brain activity, and energy expenditure in the performance of a cognitive task. Nutr Neurosci. 2019 Mar;22(3):196-206. doi: 10.1080/1028415X.2017.1360559. Epub 2017 Aug 7. PMID 28784049
- [Background] Wang YP, Gorenstein C. Psychometric properties of the Beck Depression Inventory-II: a comprehensive review. Braz J Psychiatry. 2013 Oct-Dec;35(4):416-31. doi: 10.1590/1516-4446-2012-1048. Epub 2013 Dec 23. PMID 24402217
- [Background] Thurnham DI, McCabe LD, Haldar S, Wieringa FT, Northrop-Clewes CA, McCabe GP. Adjusting plasma ferritin concentrations to remove the effects of subclinical inflammation in the assessment of iron deficiency: a meta-analysis. Am J Clin Nutr. 2010 Sep;92(3):546-55. doi: 10.3945/ajcn.2010.29284. Epub 2010 Jul 7. PMID 20610634
- [Background] Sydora BC, Fast H, Campbell S, Yuksel N, Lewis JE, Ross S. Use of the Menopause-Specific Quality of Life (MENQOL) questionnaire in research and clinical practice: a comprehensive scoping review. Menopause. 2016 Sep;23(9):1038-51. doi: 10.1097/GME.0000000000000636. PMID 27300115
- [Background] Sternberg S. High-speed scanning in human memory. Science. 1966 Aug 5;153(3736):652-4. doi: 10.1126/science.153.3736.652. PMID 5939936
- [Background] Schneider-Garces NJ, Gordon BA, Brumback-Peltz CR, Shin E, Lee Y, Sutton BP, Maclin EL, Gratton G, Fabiani M. Span, CRUNCH, and beyond: working memory capacity and the aging brain. J Cogn Neurosci. 2010 Apr;22(4):655-69. doi: 10.1162/jocn.2009.21230. PMID 19320550
- [Background] Shapley M, Blagojevic M, Jordan KP, Croft PR. The spontaneous resolution of heavy menstrual bleeding in the perimenopausal years. BJOG. 2012 Apr;119(5):545-53. doi: 10.1111/j.1471-0528.2012.03282.x. Epub 2012 Feb 8. PMID 22313942
- [Background] Scott SP, Murray-Kolb LE. Iron Status Is Associated with Performance on Executive Functioning Tasks in Nonanemic Young Women. J Nutr. 2016 Jan;146(1):30-7. doi: 10.3945/jn.115.223586. Epub 2015 Dec 9. PMID 26661838
- [Background] Santoro N. Perimenopause: From Research to Practice. J Womens Health (Larchmt). 2016 Apr;25(4):332-9. doi: 10.1089/jwh.2015.5556. Epub 2015 Dec 10. PMID 26653408
- [Background] Priest JB, Parker EO, Hiefner A, Woods SB, Roberson PNE. The Development and Validation of the FACES-IV-SF. J Marital Fam Ther. 2020 Oct;46(4):674-686. doi: 10.1111/jmft.12423. Epub 2020 Jan 31. PMID 32003487
- [Background] Namaste SM, Rohner F, Huang J, Bhushan NL, Flores-Ayala R, Kupka R, Mei Z, Rawat R, Williams AM, Raiten DJ, Northrop-Clewes CA, Suchdev PS. Adjusting ferritin concentrations for inflammation: Biomarkers Reflecting Inflammation and Nutritional Determinants of Anemia (BRINDA) project. Am J Clin Nutr. 2017 Jul;106(Suppl 1):359S-371S. doi: 10.3945/ajcn.116.141762. Epub 2017 Jun 14. PMID 28615259
- [Background] Murray-Kolb LE, Wenger MJ, Scott SP, Rhoten SE, Lung'aho MG, Haas JD. Consumption of Iron-Biofortified Beans Positively Affects Cognitive Performance in 18- to 27-Year-Old Rwandan Female College Students in an 18-Week Randomized Controlled Efficacy Trial. J Nutr. 2017 Nov;147(11):2109-2117. doi: 10.3945/jn.117.255356. Epub 2017 Sep 27. PMID 28954841
- [Background] Murray-Kolb LE, Beard JL. Iron deficiency and child and maternal health. Am J Clin Nutr. 2009 Mar;89(3):946S-950S. doi: 10.3945/ajcn.2008.26692D. Epub 2009 Jan 21. PMID 19158210
- [Background] Murray-Kolb LE, Beard JL. Iron treatment normalizes cognitive functioning in young women. Am J Clin Nutr. 2007 Mar;85(3):778-87. doi: 10.1093/ajcn/85.3.778. PMID 17344500
- [Background] Mueller ST, Piper BJ. The Psychology Experiment Building Language (PEBL) and PEBL Test Battery. J Neurosci Methods. 2014 Jan 30;222:250-9. doi: 10.1016/j.jneumeth.2013.10.024. Epub 2013 Nov 20. PMID 24269254
- [Background] Milman N, Taylor CL, Merkel J, Brannon PM. Iron status in pregnant women and women of reproductive age in Europe. Am J Clin Nutr. 2017 Dec;106(Suppl 6):1655S-1662S. doi: 10.3945/ajcn.117.156000. Epub 2017 Oct 25. PMID 29070543
- [Background] Luu P, Flaisch T, Tucker DM. Medial frontal cortex in action monitoring. J Neurosci. 2000 Jan 1;20(1):464-9. doi: 10.1523/JNEUROSCI.20-01-00464.2000. PMID 10627622
- [Background] Lozoff B, Jimenez E, Wolf AW. Long-term developmental outcome of infants with iron deficiency. N Engl J Med. 1991 Sep 5;325(10):687-94. doi: 10.1056/NEJM199109053251004. PMID 1870641
- [Background] Lewis JE, Hilditch JR, Wong CJ. Further psychometric property development of the Menopause-Specific Quality of Life questionnaire and development of a modified version, MENQOL-Intervention questionnaire. Maturitas. 2005 Mar 14;50(3):209-21. doi: 10.1016/j.maturitas.2004.06.015. PMID 15734602
- [Background] Kulasingam S, Moineddin R, Lewis JE, Tierney MC. The validity of the Menopause Specific Quality of Life Questionnaire in older women. Maturitas. 2008 Jul-Aug;60(3-4):239-43. doi: 10.1016/j.maturitas.2008.07.002. Epub 2008 Aug 29. PMID 18760553
- [Background] Jauregui-Lobera I. Iron deficiency and cognitive functions. Neuropsychiatr Dis Treat. 2014 Nov 10;10:2087-95. doi: 10.2147/NDT.S72491. eCollection 2014. PMID 25419131
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630
- [Background] Gaskell H, Derry S, Andrew Moore R, McQuay HJ. Prevalence of anaemia in older persons: systematic review. BMC Geriatr. 2008 Jan 14;8:1. doi: 10.1186/1471-2318-8-1. PMID 18194534
- [Background] Fox CJ, Mueller ST, Gray HM, Raber J, Piper BJ. Evaluation of a short-form of the Berg Card Sorting Test. PLoS One. 2013 May 14;8(5):e63885. doi: 10.1371/journal.pone.0063885. Print 2013. PMID 23691107
- [Background] Fan J, McCandliss BD, Sommer T, Raz A, Posner MI. Testing the efficiency and independence of attentional networks. J Cogn Neurosci. 2002 Apr 1;14(3):340-7. doi: 10.1162/089892902317361886. PMID 11970796
- [Background] Fallahzadeh H. Quality of life after the menopause in Iran: a population study. Qual Life Res. 2010 Aug;19(6):813-9. doi: 10.1007/s11136-010-9644-2. Epub 2010 Apr 1. PMID 20358299
- [Background] Duckitt K. Medical management of perimenopausal menorrhagia: an evidence-based approach. Menopause Int. 2007 Mar;13(1):14-8. doi: 10.1258/175404507780456782. PMID 17448262
- [Background] Delamater L, Santoro N. Management of the Perimenopause. Clin Obstet Gynecol. 2018 Sep;61(3):419-432. doi: 10.1097/GRF.0000000000000389. PMID 29952797
- [Background] Cook JD, Flowers CH, Skikne BS. The quantitative assessment of body iron. Blood. 2003 May 1;101(9):3359-64. doi: 10.1182/blood-2002-10-3071. Epub 2003 Jan 9. PMID 12521995
- [Background] Clark SF. Iron deficiency anemia. Nutr Clin Pract. 2008 Apr-May;23(2):128-41. doi: 10.1177/0884533608314536. PMID 18390780
- [Background] Camaschella C. Iron deficiency. Blood. 2019 Jan 3;133(1):30-39. doi: 10.1182/blood-2018-05-815944. Epub 2018 Nov 6. PMID 30401704
- [Background] Busti F, Campostrini N, Martinelli N, Girelli D. Iron deficiency in the elderly population, revisited in the hepcidin era. Front Pharmacol. 2014 Apr 23;5:83. doi: 10.3389/fphar.2014.00083. eCollection 2014. PMID 24795637
- [Background] Blanton CA, Green MW, Kretsch MJ. Body iron is associated with cognitive executive planning function in college women. Br J Nutr. 2013 Mar 14;109(5):906-13. doi: 10.1017/S0007114512002620. Epub 2012 Jun 7. PMID 22676919
- [Background] Bezdjian S, Baker LA, Lozano DI, Raine A. Assessing inattention and impulsivity in children during the Go/NoGo task. Br J Dev Psychol. 2009 Jun;27(Pt 2):365-83. doi: 10.1348/026151008X314919. PMID 19812711
- [Background] Beck AT, Beamesderfer A. Assessment of depression: the depression inventory. Mod Probl Pharmacopsychiatry. 1974;7(0):151-69. doi: 10.1159/000395074. No abstract available. PMID 4412100
- [Background] Beard JL, Connor JR. Iron status and neural functioning. Annu Rev Nutr. 2003;23:41-58. doi: 10.1146/annurev.nutr.23.020102.075739. Epub 2003 Apr 10. PMID 12704220
- [Background] Anderson, K., Deane, K., Lindley, D., Loucks, B., & Veach, E. (2012). The effects of time of day and practice on cognitive abilities: The PEBL Tower of London, Trail-making, and Switcher tasks (PEBL TECHNICAL REPORT 2012-04). http://sites.google.com/site/pebltechnicalreports/
- [Background] American Psychiatric Association. (2022). Diagnostic and Statistical Manual of Mental Disorders (DSM-5-TR). American Psychiatric Association Publishing. https://doi.org/10.1176/appi.books.9780890425787